CLINICAL TRIAL: NCT02075125
Title: Comparison of Prasugrel and Ticagrelor Antiplatelet Effects in Korean Patients Presenting With ST-segment Elevation Myocardial Infarction
Brief Title: Prasugrel and Ticagrelor in ST-segment Elevation Myocardial Infarction
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Enrolling participants has halted prematurely and will not resume
Sponsor: Dong-A University (Other)
Responsible Party: Principal Investigator, Moo Hyun Kim, M.D. Director, Global Clinical Trial Center. Professor, Dept. of Cardiology Dong-A Unicersity Hospital, Dong-A University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PANTASTIC
Record Dates: First submitted 2014-02-20; First posted 2014-03-03 (Estimated); Results first posted 2016-02-01 (Estimated); Last update posted 2017-08-18 (Actual); Status verified 2017-07

CONDITIONS: ST-Segment Elevation Myocardial Infarction
Keywords: Korea; Platelet inhibition; Prasugrel; Ticagrelor; ST-segment elevation myocardial infarction
MeSH Terms: conditions — ST Elevation Myocardial Infarction | interventions — Prasugrel Hydrochloride; Ticagrelor

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Prasugrel 60 mg (Experimental): Prasugrel 60 mg as loading dose and followed by 10 mg/day as maintenance dose
  Interventions: Drug: Prasugrel 60 mg
- Ticagrelor 180 mg (Experimental): Ticagrelor 180 mg as loading dose and followed by 90 mg twice a day as maintenance dose
  Interventions: Drug: Ticagrelor 180 mg

INTERVENTIONS:
Drug: Prasugrel 60 mg — Patient administer prasugrel 60 mg as loading dose followed by 10 mg/day as maintenance dose.
  Other Names: Effient 60 mg
  Arms: Prasugrel 60 mg
Drug: Ticagrelor 180 mg — Patients administer ticagrelor 180 mg as loading dose followed by 90 mg bid as maintenance dose.
  Other Names: Brilinta 180 mg
  Arms: Ticagrelor 180 mg

SUMMARY:
To compare efficacy and safety of prasugrel and ticagrelor in patients with ST-segment elevation myocardial infarction undergoing primary percutaneous coronary intervention.

DETAILED DESCRIPTION:
Prasugrel and ticagrelor are recommended in patients with ST-segment elevation myocardial infarction (STEMI) undergoing primary percutaneous coronary intervention (PCI). Both prasugrel and ticagrelor show more rapid and potent antiplatelet effect compared with clopidogrel. However, previous report comparing the efficacy and safety of prasugrel and ticagrelor in patients with STEMI of East Asian ethnicity is lacking. Therefore, the aim of this study is to compare the antiplatelet efficacy and safety using laboratory platelet function tests and clinical outcomes in patients with STEMI treated with either prasugrel or ticagrelor.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ST-segment elevation myocardial infarction
* Undergoing primary percutaneous coronary intervention
* Aged between 20 and 80 years

Exclusion Criteria:

* Previous administration of any antagonist of the platelet adenosine diphosphate (ADP) P2Y12 receptor (clopidogrel, prasugrel or ticagrelor)
* History of stroke or transient ischemic attack
* Previous gastrointestinal bleeding within 6 months, bleeding diathesis, platelet count < 100,000/mm3 or hemoglobin < 10 g/dl
* Chronic oral anticoagulation treatment
* Contraindication to the antiplatelet treatment
* Severe renal insufficiency (serum creatine>2.5 mg/dl)
* Severe hepatic dysfunction (serum liver enzyme or bilirubin>3 times normal limit)
* Sever chronic obstructive pulmonary disease (COPD) or bradycardia
* Body weight < 50 kg

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2014-01; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Moo Hyun Kim, M.D., Principal Investigator — Dong-A University Hospital, Busan, Republic of Korea
Locations (1):
- DongA University Hospital, Busan, South Korea

REFERENCES:
- [Background] Parodi G, Valenti R, Bellandi B, Migliorini A, Marcucci R, Comito V, Carrabba N, Santini A, Gensini GF, Abbate R, Antoniucci D. Comparison of prasugrel and ticagrelor loading doses in ST-segment elevation myocardial infarction patients: RAPID (Rapid Activity of Platelet Inhibitor Drugs) primary PCI study. J Am Coll Cardiol. 2013 Apr 16;61(15):1601-6. doi: 10.1016/j.jacc.2013.01.024. Epub 2013 Mar 22. PMID 23500251
- [Background] Alexopoulos D, Xanthopoulou I, Gkizas V, Kassimis G, Theodoropoulos KC, Makris G, Koutsogiannis N, Damelou A, Tsigkas G, Davlouros P, Hahalis G. Randomized assessment of ticagrelor versus prasugrel antiplatelet effects in patients with ST-segment-elevation myocardial infarction. Circ Cardiovasc Interv. 2012 Dec;5(6):797-804. doi: 10.1161/CIRCINTERVENTIONS.112.972323. Epub 2012 Nov 20. PMID 23169985
- [Derived] Lee YS, Jin CD, Kim MH, Guo LZ, Cho YR, Park K, Park JS, Park TH, Kim YD. Comparison of Prasugrel and Ticagrelor Antiplatelet Effects in Korean Patients Presenting With ST-Segment Elevation Myocardial Infarction. Circ J. 2015;79(6):1248-54. doi: 10.1253/circj.CJ-15-0270. Epub 2015 May 11. PMID 25959558

RESULTS

PARTICIPANT FLOW:
Groups:
- Prasugrel: Patient administer Prasugrel 60 mg as loading dose followed by 10 mg/day as maintenance dose.
- Ticagrelor: Patient administer Ticagrelor 180 mg as loading dose followed by 90 mg twice a day as maintenance dose.
Period: Overall Study
Arm/Group | Prasugrel | Ticagrelor
Started | 19 | 20
Completed | 19 | 19 (One patient switched to clopidogrel treatment after 18 days of ticagrelor treatment.)
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Ticagrelor: Patients administer Ticagrelor 180 mg as loading dose followed by 90 mg bid as maintenance dose.
- Total: Total of all reporting groups
Arm/Group | Prasugrel | Ticagrelor | Total
Number analyzed (Participants) | 19 | 20 | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 55 (10) | 55 (11) | 55 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 17 | 18 | 35
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 19 | 20 | 39
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 25.3 (2.7) | 24.4 (2.4) | 24.9 (2.4)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With High Platelet Reactivity
Description: Platelet reactivity were measured by VerifyNow (volumetrics accuretic，San Diego, California, USA), and vasodilator-stimulated phosphoprotein (VASP) phosphorylation P2Y12 assay (BioCytex, Marseille, France) with FACSCalibur flow cytometer (BD Biosciences, San Jose, California, USA) using. Measurement time gap +/- 12 hours were allowed. High platelet reactivity (HPR) is defined as the result of P2Y12 reaction units (PRU) >235 and platelet reactivity index (PRI) >50%.
Time Frame: 48 hours after loading dose of study drug
Population: Analysis population was performed on an intention to treat basis, descriptive analysis was performed by presenting the data as number (proportion), compared with chi-square statistics or Fisher's exact test, as appropriate.
Measure: Number; unit: participants
Arm/Group | Prasugrel | Ticagrelor
Number analyzed (Participants) | 19 | 20
participants
  PRU>235 | 0 | 0
  VASP-PRI>50% | 0 | 0

2. Secondary Outcome: Major Adverse Cardiac and Cerebrovascular Events
Description: Any major adverse cardiac and cerebrovascular event including (death, myocardial infarction, or revascularization and stroke) until day 30.
Time Frame: 30 days
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Prasugrel | Ticagrelor
Number analyzed (Participants) | 19 | 20
participants | 0 | 0

3. Secondary Outcome: Bleeding Event
Description: Any event related to bleeding including access site bleeding and peri-procedural bleeding based on Bleeding Academic Research Consortium (BARC) criteria.
Time Frame: 30 days
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Prasugrel | Ticagrelor
Number analyzed (Participants) | 19 | 20
participants | 0 | 0

4. Secondary Outcome: Adverse Drug Reaction
Description: Any adverse reaction related to study drug until 30 days after percutaneous coronary intervention.
Time Frame: 30 days
Population: Analysis population was performed on an intention to treat basis, descriptive analysis was performed by presenting the data as number, compared with chi-square statistics or Fisher's exact test, as appropriate.
Measure: Number; unit: participants
Arm/Group | Prasugrel | Ticagrelor
Number analyzed (Participants) | 19 | 20
participants | 0 | 0

5. Secondary Outcome: Pre-procedure P2Y12 Reaction Units (PRU)
Description: Platelet reactivity was measured using VerifyNow (volumetrics accuretic, San Diego, California, USA). Platelet reactivity values were presented as P2Y12 reaction units (PRU).
Time Frame: Baseline
Population: Analysis population was performed on an intention to treat basis, descriptive analysis was performed by presenting the data as median (Inter-Quartile Range).
Measure: Median (Inter-Quartile Range); unit: PRU units
Arm/Group | Prasugrel | Ticagrelor
Number analyzed (Participants) | 19 | 20
PRU units | 259 [230 to 281] | 261 [196 to 286]

6. Secondary Outcome: Number of Participants With Low Platelet Reactivity
Description: Platelet reactivity were measured using VerifyNow (volumetrics accuretic, San Diego, California, USA), and vasodilator-stimulated phosphoprotein (VASP) phosphorylation P2Y12 assay (BioCytex, Marseille, France) with FACSCalibur flow cytometer (BD Biosciences, San Jose, California, USA) using. Measurement time gap +/- 12 hours were allowed. Low platelet reactivity (LPR) is defined as the result of P2Y12 reaction units (PRU) <85 and platelet reactivity index (PRI)<16%. The PRU value for LPR, 18 patients were in prasugrel groups and 19 patients in ticagrelor groups, regarding the PRI value for LPR, 16 patients were in each groups.
Time Frame: 48 hours after loading dose of study drug
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Prasugrel | Ticagrelor
Number analyzed (Participants) | 19 | 20
participants
  PRU<85 | 18 | 19
  VASP-PRI<16% | 16 | 16

7. Secondary Outcome: Pre-procedure Platelet Reactivity Index (PRI)
Description: Platelet reactivity was measured using vasodilator-stimulated phosphoprotein (VASP) phosphorylation P2Y12 assay. Platelet reactivity values were presented as platelet reactivity index (PRI).
Time Frame: Baseline
Population: as for outcome 5
Measure: Median (Inter-Quartile Range); unit: percentage
Arm/Group | Prasugrel | Ticagrelor
Number analyzed (Participants) | 19 | 20
percentage | 51.2 [39.3 to 61.3] | 47.5 [38.4 to 50.4]

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | Prasugrel | Ticagrelor
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/20
Other Adverse Events (participants affected / at risk) | 0/19 | 0/20

LIMITATIONS AND CAVEATS:
For the present single-center pilot study, the small sample size was a major limitation, and as such was insufficiently powered to assess safety.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes